CLINICAL TRIAL: NCT02817997
Title: ACCELERATE (Advancing Castleman Care With an Electronic Longitudinal Registry, E-Repository, And Treatment/Effectiveness Research): An International Registry for Patients With Castleman Disease
Brief Title: International Registry for Patients With Castleman Disease
Acronym: ACCELERATE
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: EUSA Pharma, Inc. (Industry); Castleman Disease Collaborative Network (Other)
Responsible Party: Sponsor
Other Study IDs: 10055241; R01FD007632 (FDA)
Record Dates: First submitted 2016-06-22; First posted 2016-06-29 (Estimated); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Castleman Disease; Castleman's Disease; Giant Lymph Node Hyperplasia; Angiofollicular Lymph Hyperplasia; Angiofollicular Lymph Node Hyperplasia; Angiofollicular Lymphoid Hyperplasia; GLNH; Hyperplasia, Giant Lymph Node; Lymph Node Hyperplasia, Giant
Keywords: patient registry; ACCELERATE study; CD; MCD; iMCD; Castleman; Castleman's Disease; Angiofollicular Lymph Hyperplasia; multicentric Castleman's disease; multicentric Castleman disease
MeSH Terms: conditions — Castleman Disease; Macular dystrophy, corneal type 1; Multi-centric Castleman's Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Lymph node and/or bone marrow slides and/or tissue blocks may be sent to research team at the University of Pennsylvania to be scanned and uploaded to assist with grading likelihood of accurate diagnosis, if allowed by local regulations. Patients will be given the option to consent for lymph node and bone marrow slides collected for the registry that are determined to be unnecessary for the registry to be used for research studies, such as genomic sequencing or immunohistochemistry.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to collect clinical, laboratory, and patient survey data from patients with Castleman disease to improve understanding, diagnosis, and treatment of the disease. Funding source - FDA OOPD.

DETAILED DESCRIPTION:
This project is supported by the Castleman Disease Collaborative Network.

Visit the CDCN website at http://www.cdcn.org/accelerate to sign up for the ACCELERATE registry!

The ACCELERATE patient registry will give patients and families the opportunity to contribute their medical data to improve understanding of Castleman Disease. The patient registry will obtain real-world demographic, clinical, laboratory, and patient reported outcomes, and treatment data from 1000 patients worldwide with Castleman Disease.

This registry will help to provide important data for future Castleman Disease research studies. The patient registry helps centralize information on this rare disease, and provides researchers a way to obtain data on Castleman Disease patients. The major objectives for the registry include:

1. Improve our understanding of the natural history (signs, symptoms, laboratory values, survival data, outcome predictors), pathogenesis, and treatment of Castleman disease by collecting a standardized set of demographic and longitudinal data from CD patients,
2. Build capacity for collaboration between patients, providers, researchers, and industry by collecting clinical data and tracking the location of all available tissue samples for future studies ("virtual biorepository"), and
3. Assemble "real-world" data related to burden of disease, treatments used, tolerability, and safety data.

Individuals affected by Castleman Disease and families of deceased patients are invited to join the registry.

Patients located anywhere in the United States of America (USA), Canada, or rest of world will be able to enroll themselves directly into the registry. Participants will enroll online and be asked to provide their electronic medical records to University of Pennsylvania researchers for data extraction. All patients will also be asked to complete questionnaires every three months about their symptoms, treatments, and experiences with Castleman Disease. Complete participant information will be stored in a secure database.

Researchers who are interested in studying Castleman Disease can also request access to registry datasets.

ELIGIBILITY:
Inclusion Criteria:

* Person of any age
* Have a reference pathology report suggesting "Castleman disease" not limited to cutaneous involvement only that can be uploaded
* Be able to provide electronic informed consent, as per local regulations
* Deceased patients may also be enrolled when a reference pathology report suggesting "Castleman disease" can be supplied or when the ART is able to locate and upload such a pathology report.

Exclusion Criteria:

* Because this registry is designed to provide as wide a picture of routine clinical practice as possible, inclusion criteria are set deliberately wide and there are no exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Castleman Disease patients worldwide
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-10; Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Common Symptoms | 5 years
  There is no intervention tested in this registry. We want determine what are common symptoms are associated with Castleman Disease. We will be examining the number of instances various symptoms such as fatigue, malaise, fever are recorded in the medical records.
Common Laboratory Abnormalities | 5 years
  There is no intervention tested in this registry. We want determine what are common laboratory abnormalities associated with Castleman Disease. We will be examining the values of specific laboratory values associated with Castleman's Disease such as C-Reactive Protein (CRP), ferritin, and hemoglobin recorded in the medical records.
Treatment | 5 years
  There is no intervention tested in this registry. We want determine what are common treatments used for patients with Castleman Disease. We will be examining the number of instances specific treatments such as steroids and chemotherapy are recorded in the medical records.
Survival | 5 years
  There is no intervention tested in this registry. Distribution of time-to-event variables will be estimated using standard survival analysis methods, including Kaplan-Meier product-limit survival curves. The median time to event with 2-sided 95% confidence intervals will be estimated.
Identify patient subtypes | 4 years
  We will use data collected through this study to identify patient subgroups, particularly those that are not responsive to current treatments
Identify clinical outcome measures | 4 years
  We will use data collected through this study to determine the optimal parameters for overarching clinical outcome measures for use in future trials
Identify clinical biomarkers | 4 years
  We will use data collected through this study to identify biomarkers of treatment response

CONTACTS AND LOCATIONS:
Overall Officials: David C Fajgenbaum, MD, MBA, MSc, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified Researchers, who apply for access to the database and are subsequently approved, will be given access to a limited dataset with direct identifiers removed in an Excel compatible file format or single SAS data files. The Certification & Access Subcommittee will review applications from qualified researchers on an ongoing basis.

REFERENCES:
- [Background] Liu AY, Nabel CS, Finkelman BS, Ruth JR, Kurzrock R, van Rhee F, Krymskaya VP, Kelleher D, Rubenstein AH, Fajgenbaum DC. Idiopathic multicentric Castleman's disease: a systematic literature review. Lancet Haematol. 2016 Apr;3(4):e163-75. doi: 10.1016/S2352-3026(16)00006-5. Epub 2016 Mar 17. PMID 27063975
- [Background] Fajgenbaum DC, van Rhee F, Nabel CS. HHV-8-negative, idiopathic multicentric Castleman disease: novel insights into biology, pathogenesis, and therapy. Blood. 2014 May 8;123(19):2924-33. doi: 10.1182/blood-2013-12-545087. Epub 2014 Mar 12. PMID 24622327
- [Result] Pierson SK, Khor JS, Ziglar J, Liu A, Floess K, NaPier E, Gorzewski AM, Tamakloe MA, Powers V, Akhter F, Haljasmaa E, Jayanthan R, Rubenstein A, Repasky M, Elenitoba-Johnson K, Ruth J, Jacobs B, Streetly M, Angenendt L, Patier JL, Ferrero S, Zinzani PL, Terriou L, Casper C, Jaffe E, Hoffmann C, Oksenhendler E, Fossa A, Srkalovic G, Chadburn A, Uldrick TS, Lim M, van Rhee F, Fajgenbaum DC. ACCELERATE: A Patient-Powered Natural History Study Design Enabling Clinical and Therapeutic Discoveries in a Rare Disorder. Cell Rep Med. 2020 Dec 22;1(9):100158. doi: 10.1016/j.xcrm.2020.100158. eCollection 2020 Dec 22. PMID 33377129
- [Result] Pierson SK, Stonestrom AJ, Shilling D, Ruth J, Nabel CS, Singh A, Ren Y, Stone K, Li H, van Rhee F, Fajgenbaum DC. Plasma proteomics identifies a 'chemokine storm' in idiopathic multicentric Castleman disease. Am J Hematol. 2018 Jul;93(7):902-912. doi: 10.1002/ajh.25123. Epub 2018 May 16. PMID 29675946
- [Result] Fajgenbaum DC, Langan RA, Japp AS, Partridge HL, Pierson SK, Singh A, Arenas DJ, Ruth JR, Nabel CS, Stone K, Okumura M, Schwarer A, Jose FF, Hamerschlak N, Wertheim GB, Jordan MB, Cohen AD, Krymskaya V, Rubenstein A, Betts MR, Kambayashi T, van Rhee F, Uldrick TS. Identifying and targeting pathogenic PI3K/AKT/mTOR signaling in IL-6-blockade-refractory idiopathic multicentric Castleman disease. J Clin Invest. 2019 Aug 13;129(10):4451-4463. doi: 10.1172/JCI126091. PMID 31408438
- [Result] Arenas DJ, Floess K, Kobrin D, Pai RL, Srkalovic MB, Tamakloe MA, Rasheed R, Ziglar J, Khor J, Parente SAT, Pierson SK, Martinez D, Wertheim GB, Kambayashi T, Baur J, Teachey DT, Fajgenbaum DC. Increased mTOR activation in idiopathic multicentric Castleman disease. Blood. 2020 May 7;135(19):1673-1684. doi: 10.1182/blood.2019002792. PMID 32206779
- [Result] Pai RL, Japp AS, Gonzalez M, Rasheed RF, Okumura M, Arenas D, Pierson SK, Powers V, Layman AAK, Kao C, Hakonarson H, van Rhee F, Betts MR, Kambayashi T, Fajgenbaum DC. Type I IFN response associated with mTOR activation in the TAFRO subtype of idiopathic multicentric Castleman disease. JCI Insight. 2020 May 7;5(9):e135031. doi: 10.1172/jci.insight.135031. PMID 32376796
- [Result] van Rhee F, Oksenhendler E, Srkalovic G, Voorhees P, Lim M, Dispenzieri A, Ide M, Parente S, Schey S, Streetly M, Wong R, Wu D, Maillard I, Brandstadter J, Munshi N, Bowne W, Elenitoba-Johnson KS, Fossa A, Lechowicz MJ, Chandrakasan S, Pierson SK, Greenway A, Nasta S, Yoshizaki K, Kurzrock R, Uldrick TS, Casper C, Chadburn A, Fajgenbaum DC. International evidence-based consensus diagnostic and treatment guidelines for unicentric Castleman disease. Blood Adv. 2020 Dec 8;4(23):6039-6050. doi: 10.1182/bloodadvances.2020003334. PMID 33284946
- [Result] Koa B, Borja AJ, Aly M, Padmanabhan S, Tran J, Zhang V, Rojulpote C, Pierson SK, Tamakloe MA, Khor JS, Werner TJ, Fajgenbaum DC, Alavi A, Revheim ME. Emerging role of 18F-FDG PET/CT in Castleman disease: a review. Insights Imaging. 2021 Mar 11;12(1):35. doi: 10.1186/s13244-021-00963-1. PMID 33709329
- [Result] Nishimura Y, Fajgenbaum DC, Pierson SK, Iwaki N, Nishikori A, Kawano M, Nakamura N, Izutsu K, Takeuchi K, Nishimura MF, Maeda Y, Otsuka F, Yoshizaki K, Oksenhendler E, van Rhee F, Sato Y. Validated international definition of the thrombocytopenia, anasarca, fever, reticulin fibrosis, renal insufficiency, and organomegaly clinical subtype (TAFRO) of idiopathic multicentric Castleman disease. Am J Hematol. 2021 Oct 1;96(10):1241-1252. doi: 10.1002/ajh.26292. Epub 2021 Jul 28. PMID 34265103
- [Result] Pierson SK, Shenoy S, Oromendia AB, Gorzewski AM, Langan Pai RA, Nabel CS, Ruth JR, Parente SAT, Arenas DJ, Guilfoyle M, Reddy M, Weinblatt M, Shadick N, Bower M, Pria AD, Masaki Y, Katz L, Mezey J, Beineke P, Lee D, Tendler C, Kambayashi T, Fossa A, van Rhee F, Fajgenbaum DC. Discovery and validation of a novel subgroup and therapeutic target in idiopathic multicentric Castleman disease. Blood Adv. 2021 Sep 14;5(17):3445-3456. doi: 10.1182/bloodadvances.2020004016. PMID 34438448
- [Result] Belyaeva E, Rubenstein A, Pierson SK, Dalldorf D, Frank D, Lim MS, Fajgenbaum DC. Bone marrow findings of idiopathic Multicentric Castleman disease: A histopathologic analysis and systematic literature review. Hematol Oncol. 2022 Apr;40(2):191-201. doi: 10.1002/hon.2969. Epub 2022 Feb 18. PMID 35104370
- [Result] Phillips AD, Kakkis JJ, Tsao PY, Pierson SK, Fajgenbaum DC. Increased mTORC2 pathway activation in lymph nodes of iMCD-TAFRO. J Cell Mol Med. 2022 Jun;26(11):3147-3152. doi: 10.1111/jcmm.17251. Epub 2022 Apr 30. PMID 35488725
- [Result] Fajgenbaum DC, Pierson SK, Kanhai K, Bagg A, Alapat D, Lim MS, Lechowicz MJ, Srkalovic G, Uldrick TS, van Rhee F; ACCELERATE Registry Team. The disease course of Castleman disease patients with fatal outcomes in the ACCELERATE registry. Br J Haematol. 2022 Jul;198(2):307-316. doi: 10.1111/bjh.18214. Epub 2022 May 4. PMID 35507638
- [Result] Pierson SK, Katz L, Williams R, Mumau M, Gonzalez M, Guzman S, Rubenstein A, Oromendia AB, Beineke P, Fossa A, van Rhee F, Fajgenbaum DC. CXCL13 is a predictive biomarker in idiopathic multicentric Castleman disease. Nat Commun. 2022 Nov 24;13(1):7236. doi: 10.1038/s41467-022-34873-7. PMID 36433996
- [Result] Sarmiento Bustamante M, Shyamsundar S, Coren FR, Bagg A, Srkalovic G, Alapat D, van Rhee F, Lim MS, Lechowicz MJ, Brandstadter JD, Pierson SK, Fajgenbaum DC. Ongoing symptoms following complete surgical excision in unicentric Castleman disease. Am J Hematol. 2023 Nov;98(11):E334-E337. doi: 10.1002/ajh.27065. Epub 2023 Aug 28. No abstract available. PMID 37635628
- [Result] Pierson SK, Lim MS, Srkalovic G, Brandstadter JD, Sarmiento Bustamante M, Shyamsundar S, Mango N, Lavery C, Austin B, Alapat D, Lechowicz MJ, Bagg A, Li H, Casper C, van Rhee F, Fajgenbaum DC. Treatment consistent with idiopathic multicentric Castleman disease guidelines is associated with improved outcomes. Blood Adv. 2023 Nov 14;7(21):6652-6664. doi: 10.1182/bloodadvances.2023010745. PMID 37656441
- [Result] Mango NA, Pierson SK, Sarmiento Bustamante M, Brandstadter JD, van Rhee F, Fajgenbaum DC. Siltuximab administration results in spurious IL-6 elevation in peripheral blood. Am J Hematol. 2024 Jan;99(1):E15-E18. doi: 10.1002/ajh.27132. Epub 2023 Oct 23. No abstract available. PMID 37867418
- [Derived] Shyamsundar S, Pierson SK, Connolly CM, Teles M, Segev DL, Werbel WA, van Rhee F, Casper C, Brandstadter JD, Noy A, Fajgenbaum DC. Castleman disease patients report mild COVID-19 symptoms and mount a humoral response to SARS-CoV-2 vaccination. Blood Neoplasia. 2024 Mar;1(1):100002. doi: 10.1016/j.bneo.2024.100002. Epub 2024 Feb 15. PMID 39044861
- [Derived] Rubenstein AI, Pierson SK, Shyamsundar S, Bustamante MS, Gonzalez MV, Milller ID, Brandstadter JD, Mumau MD, Fajgenbaum DC. Immune-mediated thrombocytopenia and IL-6-mediated thrombocytosis observed in idiopathic multicentric Castleman disease. Br J Haematol. 2024 Mar;204(3):921-930. doi: 10.1111/bjh.19279. Epub 2024 Jan 2. PMID 38168727
- [Derived] Dispenzieri A, Fajgenbaum DC. Overview of Castleman disease. Blood. 2020 Apr 16;135(16):1353-1364. doi: 10.1182/blood.2019000931. PMID 32106302
- [Derived] van Rhee F, Voorhees P, Dispenzieri A, Fossa A, Srkalovic G, Ide M, Munshi N, Schey S, Streetly M, Pierson SK, Partridge HL, Mukherjee S, Shilling D, Stone K, Greenway A, Ruth J, Lechowicz MJ, Chandrakasan S, Jayanthan R, Jaffe ES, Leitch H, Pemmaraju N, Chadburn A, Lim MS, Elenitoba-Johnson KS, Krymskaya V, Goodman A, Hoffmann C, Zinzani PL, Ferrero S, Terriou L, Sato Y, Simpson D, Wong R, Rossi JF, Nasta S, Yoshizaki K, Kurzrock R, Uldrick TS, Casper C, Oksenhendler E, Fajgenbaum DC. International, evidence-based consensus treatment guidelines for idiopathic multicentric Castleman disease. Blood. 2018 Nov 15;132(20):2115-2124. doi: 10.1182/blood-2018-07-862334. Epub 2018 Sep 4. PMID 30181172
- See also: website includes information on Castleman Disease, the ACCELERATE Castleman Disease Registry, and related Castleman Disease links — http://www.cdcn.org/accelerate